CLINICAL TRIAL: NCT02821403
Title: Effects of Blue-light Blocking Lens on Visual Functions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HSEARS20140512001-03
Record Dates: First submitted 2016-06-27; First posted 2016-07-01 (Estimated); Results first posted 2017-04-07 (Actual); Last update posted 2017-04-07 (Actual); Status verified 2016-06

CONDITIONS: Effects of Blue-light Blocking Lens on Visual Functions

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Young adults (Experimental): adults without presbyopia who aged 18-35 years
  Interventions: Device: clear lens with regular coating; Device: regular coating lens with yellow tint; Device: clear lens with blue-light blocking coating
- Middle-aged adults (Experimental): adults with presbyopia who aged over 40 years
  Interventions: Device: clear lens with regular coating; Device: regular coating lens with yellow tint; Device: clear lens with blue-light blocking coating

INTERVENTIONS:
Device: clear lens with regular coating
Device: regular coating lens with yellow tint
Device: clear lens with blue-light blocking coating

SUMMARY:
Working Hypothesis: The blue-light blocking lens has no effect on the contrast sensitivity, accommodative response, color vision, and subjective grading of the quality of life and vision.

Purpose: To determine and compare the visual performances after wearing the blue-light blocking lenses in participants with and without presbyopia.

Methods: One hundred and sixty computer users (computer usage >2 hours/day) with (n=120, aged >40years) and without presbyopia (n=40, aged 18-35 years) will be recruited. Three pairs of ophthalmic lenses will be prescribed for the participants, in which one pair of them will be the blue-light blocking lenses (StressFree, Swisscoat, HK). The lenses will be used for intermediate vision (i.e., computer usage) in presbyopic group, and for distant vision in non-presbyopic group. The adaptation period for each pair of lenses will be 1 month. The pre- and post-treatment contrast sensitivity, accommodative response and color vision will be measured. The participants will also be asked to complete questionnaires about their quality of life and vision, and the performances of these ophthalmic lenses.

Significance: The blue-light blocking lens reflects the short-wavelength lights and protects the retina from "blue-light hazards"; however, blue lights are essential for various visual function and circadian rhythms. This study will evaluate the impact of the blue-light blocking lenses on visual function and quality of life, and determine whether the blue-light blocking lenses are good choices for extra ocular protection.

ELIGIBILITY:
Inclusion Criteria:

* age: 18 to 35 years OR 40 to 55 years
* daily computer usage over over 2 hours per day

Exclusion Criteria:

* visual acuity worst than 0 logMAR
* abnormal binocular and color vision
* previous history of ocular surgeries

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2014-07; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wu J, Seregard S, Algvere PV. Photochemical damage of the retina. Surv Ophthalmol. 2006 Sep-Oct;51(5):461-81. doi: 10.1016/j.survophthal.2006.06.009. PMID 16950247
- [Background] Taylor HR, Munoz B, West S, Bressler NM, Bressler SB, Rosenthal FS. Visible light and risk of age-related macular degeneration. Trans Am Ophthalmol Soc. 1990;88:163-73; discussion 173-8. PMID 2095019
- [Background] Ham WT Jr, Mueller HA, Sliney DH. Retinal sensitivity to damage from short wavelength light. Nature. 1976 Mar 11;260(5547):153-5. doi: 10.1038/260153a0. No abstract available. PMID 815821
- [Background] WALD G. THE RECEPTORS OF HUMAN COLOR VISION. Science. 1964 Sep 4;145(3636):1007-16. doi: 10.1126/science.145.3636.1007. No abstract available. PMID 14172613
- [Background] Aggarwala KR, Nowbotsing S, Kruger PB. Accommodation to monochromatic and white-light targets. Invest Ophthalmol Vis Sci. 1995 Dec;36(13):2695-705. PMID 7499092
- [Background] Kruger PB, Mathews S, Aggarwala KR, Yager D, Kruger ES. Accommodation responds to changing contrast of long, middle and short spectral-waveband components of the retinal image. Vision Res. 1995 Sep;35(17):2415-29. doi: 10.1016/0042-6989(94)00316-5. PMID 8594811
- [Background] Dijk DJ, Archer SN. Light, sleep, and circadian rhythms: together again. PLoS Biol. 2009 Jun 16;7(6):e1000145. doi: 10.1371/journal.pbio.1000145. Epub 2009 Jun 23. No abstract available. PMID 19547745
- [Background] Lockley SW, Brainard GC, Czeisler CA. High sensitivity of the human circadian melatonin rhythm to resetting by short wavelength light. J Clin Endocrinol Metab. 2003 Sep;88(9):4502-5. doi: 10.1210/jc.2003-030570. PMID 12970330
- [Derived] Leung TW, Li RW, Kee CS. Blue-Light Filtering Spectacle Lenses: Optical and Clinical Performances. PLoS One. 2017 Jan 3;12(1):e0169114. doi: 10.1371/journal.pone.0169114. eCollection 2017. PMID 28045969

RESULTS

PARTICIPANT FLOW:
Groups:
- Young Adults: adults without presbyopia who aged 18-35 years
  Three types of spectacle lenses were given to all participants: 1) clear lens with regular coating; 2) regular coating lens with yellow tint; 3) clear lens with blue-light blocking coating.
  Cross-over study design: The sequence of lens types was pseudo-randomized for each individual, i.e., participants were allocated in different sequences of lens wear by the date of admission.
- Middle-aged Adults: adults with presbyopia who aged over 40 years
  Three types of spectacle lenses were given to all participants: 1) clear lens with regular coating; 2) regular coating lens with yellow tint; 3) clear lens with blue-light blocking coating.
  Cross-over study design: The sequence of lens types was pseudo-randomized for each individual, i.e., participants were allocated in different sequences of lens wear by the date of admission.
Period: "First Intervention (1 Month)"
Arm/Group | Young Adults | Middle-aged Adults
Started | 40 | 40
Used Clear Lens | 13 | 13
Used Yellow Tinted Lens | 13 | 14
Used Blue-filtering Coated Lens | 14 | 13
Completed | 40 | 40
Not Completed | 0 | 0
Period: "Second Intervention (1 Month)"
Arm/Group | Young Adults | Middle-aged Adults
Started | 40 | 40
Used Clear Lens | 13 | 14
Used Yellow Tinted Lens | 14 | 13
Used Blue-filtering Coated Lens | 13 | 13
Completed | 40 | 40
Not Completed | 0 | 0
Period: "Third Intervention (1 Month)"
Arm/Group | Young Adults | Middle-aged Adults
Started | 40 | 40
Used Clear Lens | 14 | 13
Used Yellow Tinted Lens | 13 | 13
Used Blue-filtering Coated Lens | 13 | 14
Completed | 40 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Young Adults: adults without presbyopia who aged 18-35 years
  Three spectacle lens designs: 1) clear lens with regular coating; 2) regular coating lens with yellow tint; 3) clear lens with blue-light blocking coating: 3 types of spectacle lenses were given to all participants: 1) clear lens with regular coating; 2) regular coating lens with yellow tint; 3) clear lens with blue-light blocking coating
- Middle-aged Adults: adults with presbyopia who aged over 40 years
  Three spectacle lens designs: 1) clear lens with regular coating; 2) regular coating lens with yellow tint; 3) clear lens with blue-light blocking coating: 3 types of spectacle lenses were given to all participants: 1) clear lens with regular coating; 2) regular coating lens with yellow tint; 3) clear lens with blue-light blocking coating
- Total: Total of all reporting groups
Arm/Group | Young Adults | Middle-aged Adults | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 40 | 80
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 29 | 50
  Male | 19 | 11 | 30

OUTCOME MEASURES:

1. Primary Outcome: Contrast Sensitivity as Assessed by Mars Contrast Sensitivity Chart
Description: Contrast sensitivity was measured using the Mars contrast sensitivity letter chart (Mars Perceptrix, Chappaqua, NY). One out of three charts differing in the letter combinations was selected randomly in order to avoid memorization of the charts. The chart was placed at 50 cm with each letter subtended 2° visual angle. We followed the recording procedures as specified by the manufacturer: participants were instructed to read the letters from high to low contrasts and the test ended when two consecutive errors were made. The contrast sensitivity was scored as the log contrast sensitivity of the last correct letter minus 0.04 log unit for every prior error. The test was administered under normal (room illumination, 400 lux) and glare conditions. A brightness acuity tester set at its medium light intensity level (100 foot lamberts) simulated the glaring condition.
  A higher mean indicates improved contrast sensitivity.
Time Frame: Every 1-month interval from the date of randomization, up to 3 months
Measure: Mean (Standard Error); unit: log contrast sensitivity score
Groups:
- Young Adults: Clear Lens With Regular Coating; Young Adults: Regular Coating Lens With Yellow Tint; Young Adults: Clear Lens With Blue-light Blocking Coating: adults without presbyopia who aged 18-35 years
  Three types of spectacle lenses were given to all participants: 1) clear lens with regular coating; 2) regular coating lens with yellow tint; 3) clear lens with blue-light blocking coating.
  The sequence of lens types was pseudo-randomized for each individual, i.e., participants were allocated in different sequences of lens wear by the date of admission.
- Middle-aged Adults: Clear Lens With Regular Coating; Middle-aged Adults: Regular Coating Lens With Yellow Tint; Middle-aged Adults: Clear Lens With Blue-light Blocking Coatin: adults with presbyopia who aged over 40 years
  Three types of spectacle lenses were given to all participants: 1) clear lens with regular coating; 2) regular coating lens with yellow tint; 3) clear lens with blue-light blocking coating.
  The sequence of lens types was pseudo-randomized for each individual, i.e., participants were allocated in different sequences of lens wear by the date of admission.
Arm/Group | Young Adults: Clear Lens With Regular Coating | Young Adults: Regular Coating Lens With Yellow Tint | Young Adults: Clear Lens With Blue-light Blocking Coating | Middle-aged Adults: Clear Lens With Regular Coating | Middle-aged Adults: Regular Coating Lens With Yellow Tint | Middle-aged Adults: Clear Lens With Blue-light Blocking Coatin
Number analyzed (Participants) | 40 | 40 | 40 | 40 | 40 | 40
log contrast sensitivity score
  without glare | 1.866 (0.004) | 1.861 (0.005) | 1.856 (0.008) | 1.818 (0.014) | 1.799 (0.016) | 1.802 (0.013)
  with glare | 1.817 (0.015) | 1.802 (0.032) | 1.777 (0.035) | 1.759 (0.019) | 1.768 (0.018) | 1.785 (0.017)

2. Primary Outcome: Color Vision as Assessed by the Farnsworth Munsell 100 Hue Test
Description: The Farnsworth Munsell 100 hue test (X-Rite, USA) was used to evaluate colour vision. Each of the four trays consisted of 21 movable caps. Participants were asked to sort the randomly arranged caps following the hue order from the first to the last fixed caps. The total error score was calculated, as documented in the instruction manual, to quantify the accuracy of color discrimination.
  There are no defined endpoints to the "total error score" range.
  A lower score indicates improved color discrimination ability.
Time Frame: Every 1-month interval from the date of randomization, up to 3 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Young Adults: Clear Lens With Regular Coating | Young Adults: Regular Coating Lens With Yellow Tint | Young Adults: Clear Lens With Blue-light Blocking Coating | Middle-aged Adults: Clear Lens With Regular Coating | Middle-aged Adults: Regular Coating Lens With Yellow Tint | Middle-aged Adults: Clear Lens With Blue-light Blocking Coatin
Number analyzed (Participants) | 40 | 40 | 40 | 40 | 40 | 40
units on a scale | 30.8 (3.34) | 33.3 (3.36) | 30.1 (3.00) | 49.1 (5.49) | 54.65 (4.66) | 52.4 (5.21)

3. Secondary Outcome: Self-assessment of Lens Performance Through Questionnaire
Description: After each monthly wearing period (visits 3-5), the participants' lens performance, night vision quality and sleep quality (total 13 questions) were assessed subjectively using a questionnaire (scoring from 1 [very unsatisfactory] to 5 [very satisfactory]).
  At the end of the study, the participants were asked to choose their preferred lens type among the three pairs of lenses based on their subjective feeling of the "best lens type" (i.e., either clear lens, yellow tinted lens or blue-filtering coated lens).
  To make it clear and simple, here we only present the data on the participants choice of their preferred lens type (i.e., simply choosing the "best lens" among clear lens, yellow tinted lens or blue-filtering coated lens).
Time Frame: Every 1-month interval from the date of randomization, up to 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Young Adults | Middle-aged Adults
Number analyzed (Participants) | 40 | 40
Participants
  clear lens with regular coating | 20 | 9
  regular coating lens with yellow tint | 1 | 7
  clear lens with blue-light blocking coating | 19 | 24

ADVERSE EVENTS:
Description: There was no foreseeable safety issue and adverse effect. Serious and Other [Not Including Serious] Adverse Events were not collected/assessed.
Arm/Group | Young Adults | Middle-aged Adults
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes